CLINICAL TRIAL: NCT01995721
Title: Phase III, Single-center Clinical Trial to Evaluate the 4-valent HPV Vaccine for the Treatment and Prevention of Recurrent Respiratory Papillomatosis in Children
Brief Title: 4-valent HPV Vaccine to Treat Recurrent Respiratory Papillomatosis in Children
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Institute of Child Health, Hungary (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, dr. med habil Zsófia Meszner PhD, Professor, National Institute of Child Health, Hungary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 50934
Record Dates: First submitted 2013-11-20; First posted 2013-11-27 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Recurrent Respiratory Papillomatosis
Keywords: recurrent respiratory papillomatosis; human papillomavirus; vaccine; treatment; immunology; relapse
MeSH Terms: conditions — Recurrent respiratory papillomatosis; Recurrence | interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 4-valent HPV vaccine (Experimental): 4-valent HPV vaccine administered in months 0., 2., 6.
  Interventions: Biological: 4-valent HPV vaccine

INTERVENTIONS:
Biological: 4-valent HPV vaccine — Vaccination with 4-valent HPV vaccine in months 0., 2., 6.
  Other Names: Silgard; Gardasil

SUMMARY:
Recurrent respiratory papillomatosis in children caused by HPV 6,11 can be a life threatening condition resulting in surgical interventions. The maturing and disintegrating papillomas are the sources for the subsequent HPV relapses and immunization might slow down or even prevent this ongoing process.

After an initial immunological and ear-nose-throat (ENT) assessment children with at least 3 relapses in their patient history will be vaccinated with 4-valent HPV vaccine according to the following schedule: 0., 2., 6. months. It will be followed by an immunological and 3 ENT examinations to assess response to vaccination.

DETAILED DESCRIPTION:
1. Enrollment

   * ear-nose-throat (ENT) examination + oesophagoscopy
   * immunological assessment

     * assessment of selected humoral (antibodies) and
     * cellular immune response parameters(INF gamma and granzyme B testing)
     * in vitro and in vivo stimulation of PMBCs with the HPV-4 vaccine
2. Immunization with 4-valent HPV vaccine at 0,2,6 months
3. Follow up

   * 1 month after 3rd vaccine dose - immunological assessment (same tests as in the enrollment phase)
   * 6, 12 and 18 months after the 3rd vaccine dose - ENT + oesophagoscopy

ELIGIBILITY:
Inclusion Criteria:

* respiratory papillomatosis
* at least 3 relapses in patient history
* HPV 6 and/or 11 positive papillomas
* able to mount neutralizing antibodies

Exclusion Criteria:

* other chronic underlying condition
* other HPV type
* no antibody response

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2014-02; Primary Completion 2017-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Papilloma relapses | 18 months after the 3rd vaccine
  Number of relapses and surgical treatment needed after the 3rd vaccine dose during the 18--months follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Zsofia Meszner, MD, PhD, Principal Investigator — National Institute of Child Health
Locations (1):
- National Institute of Child Health, Budapest, Hungary